CLINICAL TRIAL: NCT04523727
Title: A 36-week, Single-Arm, Open-label Study to Evaluate the Safety and Tolerability of Ferric Citrate in Children With Hyperphosphatemia Related to Chronic Kidney Disease
Brief Title: Study to Evaluate the Safety and Tolerability of Ferric Citrate in Children With Hyperphosphatemia Related to Chronic Kidney Disease
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Keryx Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRX-0502-308
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Hyperphosphatemia Related to Chronic Kidney Disease
Keywords: hyperphosphatemia; chronic kidney disease; CKD; ferric citrate; pediatric; dialysis
MeSH Terms: conditions — Hyperphosphatemia; Renal Insufficiency, Chronic | interventions — ferric citrate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ferric citrate (Experimental): Participants aged 6 to < 17 years will receive ferric citrate for 36 weeks at a starting dose based on body weight categories.
  Interventions: Drug: ferric citrate

INTERVENTIONS:
Drug: ferric citrate — oral tablets
  Other Names: KRX-0502

SUMMARY:
This study will be conducted to assess the safety and tolerability of ferric citrate in pediatric participants with hyperphosphatemia related to chronic kidney disease (CKD).

ELIGIBILITY:
Inclusion Criteria:

* Age 6 years to <17 years at Screening.
* Weight ≥ 20 kilograms (kg) (dry weight for dialysis participants) at Screening.
* Chronic kidney disease (CKD) requiring chronic dialysis (i.e., hemodialysis or peritoneal dialysis), or CKD not on dialysis with an estimated glomerular filtration rate (eGFR) <30 milliliters per minute (mL/min)/1.73 meters squared (m^2) at Screening.
* Documented history of CKD-related hyperphosphatemia for at least 3 months prior to the screening visit.
* If participant is or is not on phosphate binder(s) at Visit 1, serum phosphorus must be:

  * 6 to <13 years: >5.8 milligrams per deciliter (mg/dL).
  * 13 to <17 years: >4.5 mg/dL.
* If participant is on phosphate binder(s) at Visit 1, and serum phosphorus is not greater than the above stated age-limit criteria, approximately 1 to 4-weeks of washout period is required and at Visit 1a or Visit 1b, serum phosphorus must be greater than the age above stated age-limit criteria.
* Transferrin saturation (TSAT) <50%.
* Serum ferritin of <650 nanograms per milliliter (ng/mL).
* Parent/legal guardian must be willing and able to give written informed consent, and child (participant) willing and able to give age-appropriate assent according to local regulatory requirements.
* Female participants of childbearing potential, defined as post menarche and not surgically sterile, must have a negative serum pregnancy test.
* Dialysis adequacy stable on current mode of dialysis prior to screening and agree to maintain dialysis prescription for the duration of the pharmacodynamic assessment period unless changes are needed for safety. A minimum dialysis adequacy (dialysis clearance of urea-dialysis time/volume of distribution of urea [Kt/V]), defined by the following:

  1. Hemodialysis adequacy: single-pool Kt/V ≥1.2 for at least 1 hemodialysis session within 2 months.
  2. Peritoneal dialysis: At least 1Kt/V reading ≥1.8 within 4 months.

Exclusion Criteria:

* Active significant GI disorder, including overt GI bleeding or active inflammatory bowel disease.
* Liver transaminases (aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) >3× the upper limit of normal at Screening.
* Unable to swallow pills, if participant requires tube feeding, ferric citrate must be taken orally and not administered via feeding tube.
* Non-renal cause of hyperphosphatemia.
* Active drug or alcohol dependence or abuse (excluding tobacco use or medicinal marijuana) within the 12 months prior to Screening or evidence of such abuse (in the opinion of the Investigator).
* Malignancy, except for participants who have been disease-free for at least 2 years after curative therapy.
* Participants with a functioning organ transplant.
* A known allergy or intolerance to ferric citrate or any of its constituents.
* Female participants who do not agree to remain abstinent or assent to use a combination of 2 of the following highly effective birth control methods for at least 28 days before the first dose, during the study (including during dose interruptions), and for at least 30 days after the last dose:

  * Barrier method of contraception: condoms (female or male) with or without a spermicidal agent, diaphragm, or cervical cap with spermicide.
  * Intrauterine device (IUD).
  * Hormone-based contraceptives which are associated with inhibition of ovulation.
* Females who are pregnant or breast-feeding other children. Participants who are being breastfed are eligible to participate in this study.
* Any other medical condition that, in the opinion of the Investigator, renders the participant unable to or unlikely to complete the trial or that would interfere with optimal participation in the trial or produce significant risk to the participant.
* The participant, in the opinion of the Investigator, is unable to adhere to the requirements of the study.
* Receipt of any investigational drug within 4 weeks before Screening.
* History of hemochromatosis or iron overload syndrome (e.g, hereditary sideroblastic anemia, thalassemia).

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2022-06-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with serious and non-serious treatment-emergent adverse events (TEAEs) including gastrointestinal (GI) AEs of special interest | up to Week 40
Number of participants with clinically significant laboratory abnormalities or changes in laboratory results | up to Week 40
Number of participants with TEAEs leading to the discontinuation of ferric citrate | up to Week 40

SECONDARY OUTCOMES:
Change from baseline in serum phosphorus to Week 12/early termination (ET) | Baseline; up to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Akebia Therapeutics Inc.
Locations (14):
- United States (14):
  - University of Alabama at Birmingham (UAB) - Children's of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - University of California, San Francisco (UCSF) - Department of Nephrology, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of South Florida, Tampa, Florida
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital - Kansas City, Kansas City, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No